CLINICAL TRIAL: NCT05418777
Title: Treatment of Pneumocystis in COPD (the TOPIC Study)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: lack of enrollment
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Matthew Sims, MD, PhD, Director Infectious Disease Research, Beaumont Health; Professor of Internal Medicine and Foundational Medical Studies, OUWB School of Medicine, Corewell Health East
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022-102
Record Dates: First submitted 2022-06-09; First posted 2022-06-14 (Actual); Results first posted 2023-11-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: COPD Exacerbation Acute
Keywords: pneumocystitis jirovecii; Chronic Obstructive Pulmonary Disease (COPD); trimethoprim-sulfamethoxazole
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Trimethoprim, Sulfamethoxazole Drug Combination; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- TMP-SMX (Experimental): Suspension with the equivalent of one DS TMP-SMX by mouth every 12 hours for 10 days
  Interventions: Drug: Trimethoprim Sulfamethoxazole
- Placebo (Placebo Comparator): Suspension with placebo by mouth every 12 hours for 10 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Trimethoprim Sulfamethoxazole — Receipt of suspension with the equivalent of one DS TMP-SMX by mouth every 12 hours for 10 days
  Other Names: Bactrim, Bactrim DS, Sulfatrim
  Arms: TMP-SMX
Drug: Placebo — Receipt of suspension with placebo by mouth every 12 hours for 10 days
  Other Names: sugar pill
  Arms: Placebo

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a progressive lung disease associated with chronic inflammation in the airways and lung, resulting in significant morbidity and mortality worldwide. Smoking is the primary risk factor for development of COPD and progression of the disease is associated with acute exacerbations of COPD (AECOPD) that can be triggered by acute bacterial or viral airway infections or can occur independently of infection. AECOPD can lead to hospitalization, progression of the disease, and mortality. COPD affects an estimated 11.7% of the world population and was the third leading cause of death worldwide in 2019.

This study is a randomized, double-blinded and placebo controlled study to determine if treating PJ in AECOPD with confirmed PJ colonization has a beneficial clinical impact. As a secondary goal of the study, it will be determined if TMP-SMX can decolonize these patients and if the decolonization is durable for at least 3 months.

The causes of progression of COPD, especially in the absence of continued tobacco use, are incompletely understood and a significant area of need. One proposed trigger for progression and increased AECOPD is colonization (presence of the organism without an actual infection) with Pneumocystis jirovecii (PJ), a fungal pathogen best known for causing pneumonia in patients with HIV or other forms of immunosuppression. It has been found to be more prevalent in those with severe COPD, particularly during AECOPD, but as a colonizer, not a cause of acute pneumonia. Several studies have linked PJ with progression of COPD, showing that PJ perpetuates an inflammatory and lung remodeling response, contributing to development of airway obstruction, emphysema and accelerating the disease course.

The aim of this study is to add trimethoprim-sulfamethoxazole (TMP-SMX) to standard of care treatment of AECOPD in patients who are colonized with PJ will improve the clinical outcome for the patient. This study is a pilot which will serve as proof of concept that screening for PJ in the AECOPD population and treating it with the commonly available, safe, and inexpensive antibiotic TMP-SMX will be an effective strategy.

DETAILED DESCRIPTION:
The current standard of care for detection of PJ has significant limitations in COPD patients. There is no reliable in vitro culture system and traditional detection methods are based on histochemical staining with direct fluorescent antibodies (DFA) that target the cyst form of the organism isolated from bronchoalveolar lavage (BAL) fluid. BAL is an invasive diagnostic procedure that often cannot be performed safely in patients with AECOPD due to associated risk of worsening respiratory failure and intubation. In non-HIV patients, PJ is at a lower bioburden and generally exists in the vegetative form rather than the cyst form. The lower PJ cyst burden leads to a lower sensitivity of DFA (20%) which specifically targets the cyst form. This in turn leads to difficulty in identifying PJ in the non-HIV population including transplant and COPD patients. This has led to a lack of clinical trials for potential therapeutic interventions targeting PJ to treat AECOPD or to prevent progression of COPD. A novel method of non-invasive sample collection of sputum analysis with the Unyvero system which is a novel nucleic acid amplification testing (NAAT) based assay demonstrated to have high sensitivity for PJ is being used to determine prevalence of PJ in the AECOPD population. The ability to routinely identify the subgroup of patients colonized with PJ among the hospitalized patients with AECOPD is a necessary step toward selection of the most appropriate potentially treatable patients to include in this pilot study designed to treat AECOPD.

Trimethoprim-sulfamethoxazole (TMP-SMX) is the standard of care for treating PJ pneumonia in HIV patients, and has been shown in prior studies to have high clinical cure rates. Our intervention is adding TMP-SMX to the treatment regimen for patients hospitalized with AECOPD and colonized with PJ. The goal of this study is to determine if treating PJ in AECOPD with confirmed PJ colonization has a beneficial clinical impact. As a secondary goal of the study, it will be determined if TMP-SMX can decolonize these patients and if the decolonization is durable for at least 3 months.

Participants will be randomized in a 1:1 ratio to one of two groups. Group #1 will receive a suspension with the equivalent of one double strength (DS) TMP-SMX by mouth every 12 hours. Group #2 will received a suspension with placebo by mouth every 12 hours. If the participant is discharged prior to completing the 10-day course of the medication, they will be sent home with the remaining days of study medication and a medication diary which will be collected at the end of therapy visit. When a patient with PJ pneumonia is hypoxic, the treatment of the PJ in addition to TMP-SMX includes steroids.

Upon consent patients will be given the COPD Assessment Test (CAT) (https://www.mdcalc.com/copd-assessment-test-cat), a validated scoring system used in COPD patients to assess progression, functional status, and effectiveness of pulmonary rehabilitation. Participants will be monitored daily while in the hospital for highest oxygen need, need for non-invasive or invasive mechanical ventilation, and adverse events, daily monitoring will be carried out by the nurse coordinator. Medications used for the treatment of COPD and antibiotics used will be collected retrospectively for each patient. If the patient remains hospitalized at end of therapy, 30 days, or 90 days then follow up will occur in the hospital. Otherwise, the patient will be asked to come to the Infectious Diseases Clinical Research Office for follow up visits at end of therapy (+0-3 days to allow for schedule issues and end of therapy falling on a weekend), 30 days +/-5 days, and 90 days +/- 10 days. A $30 stipend will be paid to the participants after each follow up visit. At the end of treatment visit, the medication diary will be collected. At each follow up visit, the nurse coordinator will review the patient's need for oxygen, their medications for the treatment of COPD, any need to see a physician or go to an urgent care or an emergency room for COPD, and any admission to the hospital for COPD. The CAT will be administered at each follow up visit. An expectorated sputum sample will be collected at each follow up visit which will be transported to the Infectious Diseases Research Laboratory for analysis; sputum samples will be processed and analyzed with the Unyvero system for presence of PJ by polymerase chain reaction (PCR).

ELIGIBILITY:
Inclusion Criteria:

* Carries the diagnosis of COPD and admitted for and admitted with AECOPD to Beaumont, Royal Oak (AECOPD requires increased cough, increased sputum production, and shortness of breath +/- increased oxygen needs from baseline)
* Able to produce a sputum sample
* Men or women, age ≥ 40 and < 90
* Previously enrolled in the EPIC Study and positive for Pneumocystis jirovecii detected in their sputum
* Currently treated with steroids
* Kidney function not severely impaired (CrCl ≥ 60)
* AST and ALT ≤5x upper limit of normal
* Willing and able to consent to the study

Exclusion Criteria:

* Current diagnosis of pneumonia or COVID-19
* Allergy or hypersensitivity to trimethoprim-sulfamethoxazole
* Current ICU admission or mechanical ventilation
* Active cancer or chemotherapy (except non-melanoma skin cancer)
* Other potentially confounding pulmonary diagnosis
* HIV, leukopenia, neutropenia, or other immunosuppressive condition or current use of immunosuppressive medications
* Presence of gastrointestinal tract abnormalities that would prevent absorption of medications
* Patients with concomitant infection requiring antibiotics active against Pneumocystis jirovecii
* Concomitant use of coumadin, phenytoin, pioglitazone, repaglinide, rosiglitazone, glipizide or glyburide
* Megaloblastic anemia due to folate deficiency
* Pregnancy
* Life expectancy less than 3 months

Ages: 40 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-09-28 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2022-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Sims, MD, PhD, Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TMP-SMX | Placebo
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants were enrolled and randomized to the placebo arm
Groups:
- Total: Total of all reporting groups
Arm/Group | TMP-SMX | Placebo | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Continuous [Mean (Full Range); unit: years] | 64 [64 to 64] |  | 64 [64 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 1
  Male | 0 |  | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in the COPD Assessment Test
Description: Change in total score on the COPD Assessment Test (CAT); the test has a score of 0 (minimum) - 40 (maximum); a lower score means a better outcomes and a higher score means a worse outcome. Negative numbers indicate improvement of condition. Positive numbers indicate worsening of condition.
Time Frame: Baseline to 3 months
Population: No participants were enrolled and randomized to the placebo arm
Measure: Mean (Standard Deviation); unit: number on a scale
Arm/Group | TMP-SMX | Placebo
Number analyzed (Participants) | 1 | 0
number on a scale
  Baseline to Day 10 | -10 (0) |
  Baseline to Day 30 | -6 (0) |
  Baseline to Day 90 | -2 (0) |

2. Secondary Outcome: Length of Stay for Current AECOPD
Description: Length of stay in the hospital for index exacerbation measured in days
Time Frame: up to 3 months
Population: No participants were enrolled and randomized to the placebo arm
Measure: Mean (Standard Deviation); unit: numbers of days
Arm/Group | TMP-SMX | Placebo
Number analyzed (Participants) | 1 | 0
numbers of days | 5 (0) |

3. Secondary Outcome: Time to Return to Baseline Oxygen for the Current AECOPD
Description: Time to return to baseline oxygenation for the index exacerbation measured in days
Time Frame: up to 3 months
Population: No participants were enrolled and randomized to the placebo arm
Measure: Mean (Standard Deviation); unit: days
Arm/Group | TMP-SMX | Placebo
Number analyzed (Participants) | 1 | 0
days | 0 (0) |

4. Secondary Outcome: Interval Between Exacerbations of COPD
Description: Time between exacerbation of COPD measured in days
Time Frame: up to 3 months
Population: No participants were enrolled and randomized to the placebo arm
Measure: Mean (Standard Deviation); unit: days
Arm/Group | TMP-SMX | Placebo
Number analyzed (Participants) | 1 | 0
days
  Baseline to 1st exacerbation | 33 (0) |
  1st exacerbation to 2nd exacerbation | 7 (0) |

5. Secondary Outcome: Interval Between Hospital Admissions
Description: Time before next admission to the hospital measured in days
Time Frame: up to 3 months
Population: No participants were enrolled and randomized to the placebo arm
Measure: Mean (Standard Deviation); unit: days
Arm/Group | TMP-SMX | Placebo
Number analyzed (Participants) | 1 | 0
days | 40 (0) |

6. Secondary Outcome: Number of Urgent Care Visits (Total)
Description: Total number of urgent care visits following the index exacerbation
Time Frame: up to 3 months
Population: No participants were enrolled and randomized to the placebo arm
Measure: Mean (Standard Deviation); unit: number of visits
Arm/Group | TMP-SMX | Placebo
Number analyzed (Participants) | 1 | 0
number of visits | 0 (0) |

7. Secondary Outcome: Number of Urgent Care Visits (Related to COPD)
Description: Number of urgent care visits related to COPD following the index exacerbation
Time Frame: up to 3 months
Population: No participants were enrolled and randomized to the placebo arm
Measure: Mean (Standard Deviation); unit: number of visits
Arm/Group | TMP-SMX | Placebo
Number analyzed (Participants) | 1 | 0
number of visits | 0 (0) |

8. Secondary Outcome: Number of Hospital Admissions (Total)
Description: Total number of hospital admissions following the index exacerbation
Time Frame: up to 3 months
Population: No participants were enrolled and randomized to the placebo arm
Measure: Mean (Standard Deviation); unit: number of visits
Arm/Group | TMP-SMX | Placebo
Number analyzed (Participants) | 1 | 0
number of visits | 1 (0) |

9. Secondary Outcome: Number of Hospital Admissions (Related to COPD)
Description: Number of hospital admissions related to COPD following the index exacerbation
Time Frame: up to 3 months
Population: No participants were enrolled and randomized to the placebo arm
Measure: Mean (Standard Deviation); unit: number of visits
Arm/Group | TMP-SMX | Placebo
Number analyzed (Participants) | 1 | 0
number of visits | 1 (0) |

10. Secondary Outcome: Clearance of PJ From Treated Patients
Description: Number of patients that show clearance of PJ
Time Frame: up to 3 months
Population: No participants were enrolled and randomized to the placebo arm
Measure: Count of Participants; unit: Participants
Arm/Group | TMP-SMX | Placebo
Number analyzed (Participants) | 1 | 0
Participants | 1 |

11. Secondary Outcome: Durability of Clearance of PJ From Treated Patients
Description: Number of patients who cleared PJ and did not show re-colonization with pathogen
Time Frame: up to 3 months
Population: No participants were enrolled and randomized to the placebo arm
Measure: Count of Participants; unit: Participants
Arm/Group | TMP-SMX | Placebo
Number analyzed (Participants) | 1 | 0
Participants | 1 |

12. Secondary Outcome: Need for Medications to Treat COPD
Description: Number of medications used to treat COPD
Time Frame: up to 3 months
Population: No participants were enrolled and randomized to the placebo arm
Measure: Mean (Standard Deviation); unit: number of medications
Arm/Group | TMP-SMX | Placebo
Number analyzed (Participants) | 1 | 0
number of medications | 5 (0) |

13. Secondary Outcome: Need for Mechanical Ventilation
Description: Number of participants who required mechanical ventilation
Time Frame: up to 3 months
Population: No participants were enrolled and randomized to the placebo arm
Measure: Count of Participants; unit: Participants
Arm/Group | TMP-SMX | Placebo
Number analyzed (Participants) | 1 | 0
Participants | 0 |

14. Secondary Outcome: Mortality
Description: Number of participants who died
Time Frame: up to 3 months
Population: No participants were enrolled and randomized to the placebo arm
Measure: Count of Participants; unit: Participants
Arm/Group | TMP-SMX | Placebo
Number analyzed (Participants) | 1 | 0
Participants | 0 |

ADVERSE EVENTS:
Time Frame: 3 months
Description: No participants were enrolled and randomized to the placebo arm
Arm/Group | TMP-SMX | Placebo
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TMP-SMX (N=1) | Placebo (N=0)
Candida Vaginitis (Infections and infestations) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Study was terminated due to high screen failure rate leading to low enrollment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-08): https://cdn.clinicaltrials.gov/large-docs/77/NCT05418777/Prot_SAP_000.pdf